CLINICAL TRIAL: NCT02296476
Title: A Phase IIa Trial With Dose Optimization of OTX015, a Small Molecule Inhibitor of the Bromodomain and Extra-terminal (BET) Proteins, in Recurrent Glioblastoma Multiforme (GBM) Patients
Brief Title: A Dose-finding Study of Birabresib (MK-8628) in Participants With Recurrent Glioblastoma Multiforme (MK-8628-002)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to lack of clinical activity and not due to safety reasons.
Sponsor: Oncoethix GmbH, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8628-002; OTX015_107 (Other: OncoEthix Protocol Number); MK-8628-002 (Other: Merck Protocol Number); 2014-001469-28 (EudraCT Number)
Record Dates: First submitted 2014-10-03; First posted 2014-11-20 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — OTX015

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Birabresib 80 mg (Experimental): Participants received 80 mg of oral birabresib administered once daily (in a fasted state) every day in a 28-day cycle for up to 6 cycles.
  Interventions: Drug: Birabresib
- Birabresib 120 mg (Experimental): Participants received 120 mg of oral birabresib administered once daily (in a fasted state) every day in a 28-day cycle for up to 6 cycles.
  Interventions: Drug: Birabresib
- Birabresib 160 mg (Experimental): Participants received 160 mg of oral birabresib administered once daily (in a fasted state) every day in a 28-day cycle for up to 6 cycles.
  Interventions: Drug: Birabresib

INTERVENTIONS:
Drug: Birabresib — Administered orally in a fasted state once daily.
  Other Names: OTX015; MK-8628

SUMMARY:
A study of single-agent birabresib (MK-8628) (formerly known as OTX015) in recurrent GBM after standard front-line therapy failure.

The first phase of the study (dose escalation) will determine the maximum tolerated dose (MTD). MTD assessment will be based using dose-limiting toxicities (DLTs) observed during the first 28 days of treatment.

The second phase of the study (expansion cohort) will assess efficacy as measured by the progression-free survival rate at 6 months (PFS-6) as determined by an independent central review committee.

ELIGIBILITY:
Inclusion Criteria:

* Has signed informed consent obtained prior to initiation of any study-specific procedures and treatment. Participants registered for this trial must be treated and followed at the participating centers
* Has a histologically confirmed diagnosis of de novo glioblastoma multiforme (World Health Organization grade IV astrocytoma) with unequivocal tumor recurrence by magnetic resonance imaging (MRI) scan (performed on a stable steroid dosage received for at least 5 days) following front-line treatment with surgical resection, cranial radiotherapy and temozolomid. Participants who do not undergo surgical resection as part of front-line therapy due to anatomical location based on neurosurgeon's assessment will be permitted if a confirmatory tumor biopsy was performed
* Has at least one measurable and/or non-measurable lesion as per Response Assessment in Neuro-Oncology (RANO) criteria (Wen et al., 2010)
* Is at least 18 years old
* Has a life expectancy >3 months;
* Has a Karnofsky performance status (KPS) ≥70%
* Has adequate bone marrow reserve, renal and liver function as demonstrated by the following: absolute neutrophil count ≥1.5 x109/L; platelet count ≥150 x109/L; hemoglobin ≥10 g/dL; creatinine 2 x the upper limit of normal (ULN) or calculated creatinine clearance ≥30 mL/min (Cockroft and Gault formula or Modification of Diet in Renal Disease [MDRD] formula for participants aged >65 years); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x ULN, and total bilirubin ≤ULN
* Has an interval of ≥2 weeks since surgical resection, ≥4 weeks since chemotherapy (≥6 weeks for nitrosoureas), and ≥12 weeks since radiotherapy completion when starting study treatment. Participants with recent tumor resection must have an MRI within 48 hours post-surgery
* Has archived tumor pathology specimen (paraffin-embedded or frozen block)

Exclusion Criteria:

* Has had prior antineoplastic treatment for recurrent disease including vascular endothelial growth factor (VEGF)/vascular endothelial growth factor receptor (VEGFR) inhibitors and cytotoxic agents
* Is unable to undergo MRI because of non-compatible devices
* Is unable to swallow oral medications or presence of a gastrointestinal disorder (e.g. malabsorption, resection) deemed to jeopardize intestinal absorption
* Has persistent grade >1 clinically significant toxicities related to prior antineoplastic therapies
* Has a history of prior or concomitant malignancies within 5 years of study entry (other than excised non-melanoma skin cancer or cured in situ cervical carcinoma). Male participants with concurrent controlled hormone dependent prostate cancer are allowed
* Has other serious illness or medical conditions which in the investigator's opinion could hamper understanding of the study by the participant, the participant's compliance to study treatment, participant's safety, or interpretation of study results. These include (but are not restricted to) existence of significant neurologic or psychiatric disorders impairing the ability to obtain consent, uncontrolled infection and known HIV positivity
* Is taking enzyme-inducing antiepileptic drug (EIAED)
* Is taking strong CYP3A4 interacting drugs
* Is participating in another clinical trial or treatment with any investigational drug within 4 weeks prior to first study treatment administration, or 5 half-lives of previously administered drugs, whichever is longer
* Is pregnant or breast feeding
* Is not using effective contraception while on study treatment if a participant of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10-29 (Actual); Primary Completion 2015-10-20 (Actual); Study Completion 2015-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants had a confirmed diagnosis of de novo glioblastoma multiforme (World Health Organization grade IV astrocytoma) with tumor recurrence following standard front-line treatment with surgery, cranial radiotherapy and temozolomide. Other inclusion and exclusion criteria applied.
Groups:
- MK-8628 80 mg: Participants received 80 mg of oral MK-8628 administered once daily (in a fasted state) every day in a 28-day cycle for up to 6 cycles.
- MK-8628 120 mg: Participants received 120 mg of oral MK-8628 administered once daily (in a fasted state) every day in a 28-day cycle for up to 6 cycles.
- MK-8628 160 mg: Participants received 160 mg of oral MK-8628 administered once daily (in a fasted state) every day in a 28-day cycle for up to 6 cycles.
Period: Overall Study
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Started | 6 | 4 | 2
Completed | 0 | 0 | 0
Not Completed | 6 | 4 | 2
Not completed — Disease Progression | 6 | 4 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg | Total
Number analyzed (Participants) | 6 | 4 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (14.2) | 55.8 (11.2) | 54.5 (21.9) | 52.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 4 | 4 | 2 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at 6 Months
Description: Progression-free survival was the time from the start of study treatment to the date of clinical or radiographic evidence of progressive disease according to Response Assessment in Neuro-Oncology (RANO) 2010 criteria or death. Progression, as assessed by RANO 2010, was defined as a ≥25% increase in sum of the products of perpendicular diameters of enhancing lesions; any new lesion; or clinical deterioration. PFS at 6 months was measured as the percentage of participants who were alive and progression-free at Month 6. PFS at 6 months was calculated for all participants who were actively enrolled in the study at the 6-month time point.
Time Frame: Month 6
Population: All participants who received at least 2 complete cycles (8 weeks) of treatment and had a baseline assessment and 1 on-study magnetic resonance imaging (MRI). Since no participants reached the 6-month time point in the study, PFS at 6 months could not be calculated.
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the number of participants in the analysis population who experienced a Complete Response (CR: complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks; no new lesions; no corticosteroids; and stable or improved clinically) or a Partial Response (PR: ≥50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; no new lesions; stable or reduced corticosteroid dose; and stable or improved clinically) and was assessed using RANO 2010.
Time Frame: Up to 6 Months
Population: All participants who received at least 2 complete cycles (8 weeks) of treatment and had a baseline assessment and 1 on-study MRI or had discontinued early due to disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
Participants | 0 | 0 | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was the time from the first documented CR (complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks; no new lesions; no corticosteroids; and stable or improved clinically)or PR (≥50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; no new lesions; stable or reduced corticosteroid dose; and stable or improved clinically), as assessed by RANO 2010, until documentation of disease progression, or the date of the last tumor assessment (if there was no documented progression), or the last tumor assessment before the start of further antitumor therapy. DOR was calculated for all participants who experienced a CR or PR.
Time Frame: Up to 6 Months
Population: All participants who received at least 2 complete cycles (8 weeks) of treatment and had a baseline assessment and 1 on-study MRI or had discontinued early due to disease progression. Since no participants experienced a CR or PR, DOR could not be calculated.
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Overall Survival (OS)
Description: OS was the time from the start of study treatment to the date of death. Participants were to be censored at their last contact if they were still alive at the cut-off date. OS was calculated for all participants who did not discontinue from the study due to disease progression.
Time Frame: Up to 6 Months
Population: All participants who received at least 2 complete cycles (8 weeks) of treatment and had a baseline assessment and 1 on-study MRI or had discontinued early due to disease progression. Since all participants discontinued the study due to disease progression, OS could not be calculated.
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was the time from the start of study treatment to the date of clinical or radiographic evidence of progressive disease according to RANO 2010 criteria or death. Progression, as assessed by RANO 2010, was defined as a ≥25% increase in sum of the products of perpendicular diameters of enhancing lesions; any new lesion; or clinical deterioration. PFS was measured as the number of participants who were alive and progression-free for up to 6 months.
Time Frame: Up to 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. The number of participants who experienced at least one AE is presented.
Time Frame: Up to 6 Months
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
Participants | 6 | 4 | 2

7. Secondary Outcome: Number of Participants Who Experienced at Least One Toxicity Grade 3-5 AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. The number of participants who experienced ≥1 Grade 3-5 AE per National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.03 criteria is presented. Grade 3 was classified as severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care; Grade 4 was classified as potentially life-threatening or disabling; and Grade 5 was an AE resulting in death.
Time Frame: Up to 6 Months
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
Participants | 3 | 1 | 2

8. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to 6 Months
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT) During Cycle 1
Description: A DLT was defined as any of the following toxicities that were considered by the investigator to be related to MK-8628: Hematologic toxicity: Grade 4 hematologic toxicity or febrile neutropenia, Grade 3 neutropenia with infection, Grade 3 thrombocytopenia with bleeding or lasting >7 days; Non-hematologic toxicity: Grade 3 or 4 non-hematologic toxicity (regardless of duration) unless it was not optimally managed with supportive care, Grade 3 or 4 laboratory abnormality lasting >7 days, or intolerable Grade 2 non-hematologic toxicity resulting in study treatment discontinuation or delay >7 days with or without dose reduction.
Time Frame: Up to Cycle 1 (Up to 28 days)
Population: All participants who received at least 21 days of the planned dose of study drug during the first 28-day cycle or experienced a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
Participants | 1 | 0 | 2

10. Secondary Outcome: Observed Maximum Concentration (Cmax) of MK-8628
Description: Blood samples were obtained at specified time points for the pharmacokinetic (PK) analysis of Cmax of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry and Cmax was calculated using the nonlinear mixed-effects modelling software program Monolix version 4.3.2s. The Cmax of MK-8628 after oral administration is presented.
Time Frame: Day 1: Predose and 0.25, 1, 2, 3, 7, and 8 hours postdose
Population: All participants who received MK-8628 and had blood samples drawn for PK analyses.
Measure: Mean (Standard Deviation); unit: μg/Liter
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
μg/Liter | 1022 (377) | 1138 (527) | 2725 (NA) — Standard deviation could not be estimated for 2 participants.

11. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-8628
Description: Blood samples were obtained at specified time points for the PK analysis of Tmax of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry and Tmax was calculated using the nonlinear mixed-effects modelling software program Monolix version 4.3.2s. The Tmax of MK-8628 after oral administration is presented.
Time Frame: Day 1: Predose and 0.25, 1, 2, 3, 7, and 8 hours postdose
Population: All participants who received MK-8628 and had blood samples drawn for PK analyses.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
hours | 1.7 (0.498) | 2.50 (0.572) | 2.04 (NA) — Standard deviation could not be estimated for 2 participants.

12. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of MK-8628
Description: Blood samples were obtained at specified time points for the PK analysis of t1/2 of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry and t1/2 was calculated using the nonlinear mixed-effects modelling software program Monolix version 4.3.2s. The t1/2 of MK-8628 after oral administration is presented.
Time Frame: Day 1: Predose and 0.25, 1, 2, 3, 7, and 8 hours
Population: All participants who received MK-8628 and had blood samples drawn for PK analyses.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
hours | 3.78 (0.366) | 3.74 (0.431) | 3.50 (NA) — Standard deviation could not be estimated for 2 participants.

13. Secondary Outcome: Apparent Total Body Clearance (Cl/F) of MK-8628
Description: Blood samples were obtained at specified time points for the PK analysis of Cl/F of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry and Cl/F was calculated using the nonlinear mixed-effects modelling software program Monolix version 4.3.2s. The Cl/F of MK-8628 after oral administration is presented.
Time Frame: Day 1: Predose and 0.25, 1, 2, 3, 7, and 8 hours
Population: All participants who received MK-8628 and had blood samples drawn for PK analyses.
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
Liters/hour | 10.4 (2.19) | 13.0 (4.03) | 7.75 (NA) — Standard deviation could not be estimated for 2 participants.

14. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of MK-8628
Description: Blood samples were obtained at specified time points for the PK analysis of Vz/F of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry and Vz/F was calculated using the nonlinear mixed-effects modelling software program Monolix version 4.3.2s. The Vz/F of MK-8628 after oral administration is presented.
Time Frame: Day 1: Predose and 0.25, 1, 2, 3, 7, and 8 hours
Population: All participants who received MK-8628 and had blood samples drawn for PK analyses.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
Liters | 56.3 (9.73) | 70.3 (24.1) | 39.3 (NA) — Standard deviation could not be estimated for 2 participants.

15. Secondary Outcome: Observed Minimum Concentration (Cmin) of MK-8628
Description: Blood samples were obtained at specified time points for the PK analysis of Cmin of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry. A single Cmin value for MK-8628 was estimated using dose and steady-state predose concentrations of MK-8628 on Days 29 and 57. The Cmin of MK-8628 after oral administration is presented.
Time Frame: Predose on Days 29 and 57
Population: All participants who received MK-8628 and had predose blood samples drawn on Days 29 and 57 for steady state MK-8628 concentration. Participants in the 160 mg dose group were not analyzed for Cmin because they discontinued before Day 29.
Measure: Mean (Standard Deviation); unit: μg/Liter
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 1 | 3 | 0
μg/Liter | 85.4 (NA) — Not calculated on only 1 participant | 54.1 (35.4) |

16. Secondary Outcome: Area Under the Concentration-time Curve of MK-8628 From Time 0 to Infinity (AUC 0-∞)
Description: Blood samples were obtained at specified time points for the PK analysis of AUC 0-∞ of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry. The AUC 0-∞ was estimated indirectly using the dose and CL/F values. The AUC 0-∞ of MK-8628 after oral administration is presented.
Time Frame: Day 1: Predose and 0.25, 1, 2, 3, 7, and 8 hours
Population: All participants who received MK-8628 and had blood samples drawn for PK analyses.
Measure: Mean (Standard Deviation); unit: μg•hours/Liter
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
Number analyzed (Participants) | 6 | 4 | 2
μg•hours/Liter | 8028 (2083) | 10200 (4312) | 20700 (NA) — Standard deviation could not be estimated for 2 participants.

ADVERSE EVENTS:
Time Frame: Up to 6 months (Day 1 through 28 of each treatment cycle for a maximum of 6 treatment cycles)
Description: The Safety Population consisted of all participants who received at least one dose of study treatment.
Arm/Group | MK-8628 80 mg | MK-8628 120 mg | MK-8628 160 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/4 | 2/2
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8628 80 mg (N=6) | MK-8628 120 mg (N=4) | MK-8628 160 mg (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8628 80 mg (N=6) | MK-8628 120 mg (N=4) | MK-8628 160 mg (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular icterus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (3) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (5) | 2 (2) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 2 (2) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated 31-Aug-2015 because no clinical activity was detected. The study was not terminated due to safety reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the opportunity to review proposed publications regarding this trial 45 days prior to submission for publication. Publication can be withheld an additional 90 days to allow for filing a patent or taking other measures to establish and preserve proprietary rights. Publication of the results of the study shall be made only as part of a publication of the results obtained by all sites performing the study.